CLINICAL TRIAL: NCT01256307
Title: Effects of an Individualized Training Program on Severity Markers of Obstructives Sleep Apnea/Hypopnea Syndrome (OSAS)
Acronym: REEVASAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8508
Record Dates: First submitted 2010-10-28; First posted 2010-12-08 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Sleep Apnea, Obstructive; Exercise Training Therapy
Keywords: Obstructive Sleep Apnea/Hypopnea Syndrome; Exercise training program; Inflammation; Oxidative Stress; Insulin resistance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- training group (Experimental): training and educational program
  Interventions: Other: training and educational program
- control group (Other)
  Interventions: Other: educational program

INTERVENTIONS:
Other: training and educational program — 8 weeks
  Arms: training group
Other: educational program — 8 weeks
  Arms: control group

SUMMARY:
There are two types of treatments depending on the severity of Obstructive Sleep Apnea/Hypopnea Syndrome (OSAS): - for the treatment of severe (AHI> 30/h), the standard treatment is Continuous Positive Airway Pressure (CPAP). If it proved effective in reducing excessive daytime sleepiness and associated cardiovascular risk, compliance of patients 4 years of treatment falls below 70%. - Treatment of moderate (AHI between 15 and 30/h), lifestyle measures, the bracing of mandibular advancement and / or possibly the head and neck surgery can be proposed. These treatments include side effects and their effectiveness is very controversial.Il therefore seemed interesting to test the impact of physical activity through a standardized training program to re personal effort on the development and improvement of OSAS patients with a sedentary moderate to severe OSAS (AHI between 15 and 40 / h) The main assumption is that the ESR could eventually delay the initiation of treatment with CPAP in severe OSAS or an alternative therapeutic relevance in the moderate OSAS and severe in patients who can not tolerate conventional treatment(CSF). The main objective of this biomedical research is to evaluate the effects of a program of REE in ambulatory index of hourly apneas / hypopneas (AHI = marker of severity of OSAS) .- objectives specify 2AIR effects of REE on the quality of sleep (TxSLP) and daytime symptoms (EDS objective fatigue) on the one hand and the other on the metabolism (OV, SM, IR) and markers of LCR (inflammation, oxidative stress , endothelial function).

ELIGIBILITY:
Inclusion Criteria:

* Presence of an OSAS
* Apnea Hypopnea Index between 15 and 45/h
* Sedentary subjects (Voorips Activity questionnaire)
* IMC<40

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change delta index of hourly apneas/hypopneas at eight weeks after inclusion | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

REFERENCES:
- [Derived] Bughin F, Desplan M, Mestejanot C, Picot MC, Roubille F, Jaffuel D, Mercier J, Jaussent I, Dauvilliers Y. Effects of an individualized exercise training program on severity markers of obstructive sleep apnea syndrome: a randomised controlled trial. Sleep Med. 2020 Jun;70:33-42. doi: 10.1016/j.sleep.2020.02.008. Epub 2020 Feb 18. PMID 32193052